CLINICAL TRIAL: NCT02335827
Title: Irreversible Electroporation (IRE) for Unresectable Renal Tumors: Phase I and Phase II Clinical Trial
Brief Title: Irreversible Electroporation(IRE) For Unresectable Renal Tumors
Acronym: IRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRE-001
Record Dates: First submitted 2015-01-02; First posted 2015-01-12 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2020-06

CONDITIONS: Renal Tumor
Keywords: irreversible electroporation; renal tumor
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Electroporation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): irreversible electroporation with voltage in level A for renal tumors
  Interventions: Procedure: irreversible electroporation
- Group B (Experimental): irreversible electroporation with voltage in level B for renal tumors
  Interventions: Procedure: irreversible electroporation
- Group C (Experimental): irreversible electroporation with voltage in level C for renal tumors
  Interventions: Procedure: irreversible electroporation

INTERVENTIONS:
Procedure: irreversible electroporation — Percutaneous (CT-guided and/or US-guided) or open IRE with voltage in level B for renal tumors

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of irreversible electroporation (IRE) for unresectable renal tumors.

DETAILED DESCRIPTION:
By enrolling patients with renal tumors adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of percutaneous or intraoperative IRE for renal tumors .

ELIGIBILITY:
Inclusion Criteria:

* unresectable kidney tumors
* patients refused surgical therapy
* Karnofsky-index >70%
* Age ≥ 18 and ≤ 80 years
* life expectancy ≥ 12 month
* compliance of the patient taking part in a study
* informed consent

Exclusion Criteria:

* violation against one or more inclusion criteria
* an estimated glomerular filtration rate (eGFR) of < 30 mL/min/1.73 m2
* QT-interval >550 ms or cardiac arrhythmias or condition after myocardial infarction, that make an ECG-synchronisation unfeasible
* active infection or severe health interference, that make taking part in a study unfeasible
* pregnancy, lactation period
* general contraindications for anesthesia, endotracheal anesthesia and muscle relaxation
* psychiatric disorders that make taking part in a study or giving informed consent unfeasible
* haemorrhage, impossible intermission of taking blood thinner, untreatable thrombophilia
* thromboplastin time ≤50 %, thrombocytes ≤50 Gpt/L; partial thromboplastin time >50
* untreated urinary retention
* severe hepatic dysfunction
* any other clinically important renal, hematological, metabolic, neurological, gastrointestinal, hepatic or pulmonary disorders or dysfunctions preventing study participation (investigator's assessment)
* taking part in another clinical study for renal tumor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
adverse effects | 1 month
  adverse effects measured by such as abdominal bleeding, continuous abdominal pain, renal failure, et al.
Quality of Life (QoL) | 2 months
  Quality of Life assessed as WHOQOL-BREF.
procedural compliance | 3 months
  compliance will be analyzed by 3 months of follow-up post procedure.

SECONDARY OUTCOMES:
Recurrence rate | 12 months
  efficacy assessment by percentage of lesions that show no sign of recurrence 12 months after the initial IRE procedure) of IRE for renal tumor via cross-sectional imaging and pathological examination.
Voltage (A minimum and maximum range of voltage for safe and effective IRE) | 3 months
  A minimum and maximum range of voltage for safe and effective IRE will be analyzed for optimal choice.

OTHER OUTCOMES:
Progress free disease (PFS) | 12 months
  Patients will be followed for 12 months after IRE for PFS assessing.
Overall survival (OS) | 36 months
  Patients will be followed for 36 months after IRE for OS analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PHD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Fuda Cancer Hospital, Guangzhou, Guangdong, China